CLINICAL TRIAL: NCT01268826
Title: DESHYDRAT : Assessment of the Prevalence of Dehydration Among 9 to 11 Year-old Children.
Acronym: DESHYDRAT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Direction of Clinical Research, Rennes University Hospital
Other Study IDs: 2010-A00482-37; LOC/10-04 - DESHYDRAT (Other: Rennes University Hospital); B100522-20 (Other: AFSSAPS)
Record Dates: First submitted 2010-07-20; First posted 2010-12-31 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dosage of the urinary osmolality: dosage of the urinary osmolality

SUMMARY:
The aim of the study is to determinate the prevalence of moderate dehydration among children aged 9 to 11 who are going to school.

DETAILED DESCRIPTION:
Many children have a limited caloric intake at the breakfast with a limited amount of water intake. There is no data about the prevalence of dehydration in children who are regularly going to school in France.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child aged 9 to 11 years old.

Exclusion Criteria:

* Individual with illness
* Individual with past history of gut or metabolic diseases
* Past history of renal disease.
* Child whom parents decline to participate

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 500 children aged 9-11
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of dehydration (as defined as urinary osmolality > 800 mOsmol/l) Osmolality is measured by freezing point depression | Day 1
  Prevalence of dehydration (as defined as urinary osmolality > 800 mOsmol/l) Osmolality is measured by freezing point depression

SECONDARY OUTCOMES:
Amount of water intake at breakfast | Day 1
  To determine whether urinary osmolality is correlated to total water intake at breakfast
Total energy and nutrient intake | Day 1
  To determine whether urinary osmolality is correlated to nutrient and energy intake at breakfast.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bonnet, MD, PU-PH, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France